CLINICAL TRIAL: NCT00436501
Title: Phase I/II and Pharmacokinetic Study of Docetaxel Plus VEGF Trap (AVE0005, NSC# 724770) in Patients With Recurrent Ovarian, Primary Peritoneal, and Fallopian Tube Cancer
Brief Title: VEGF Trap and Docetaxel in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00218; 2006-0329; P50CA083639 (NIH); NCT00427518 (obsolete NCT alias)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Fallopian Tube Cancer; Malignant Tumor of Peritoneum; Recurrent Ovarian Epithelial Cancer
Keywords: primary peritoneal cavity cancer; Ovarian Epithelial Cancer; Peritoneal Cancer; Fallopian Tube Cancer; VEGF Trap; aflibercept; vascular endothelial growth factor trap; Zaltrap; docetaxel; RP 56976; Taxotere; TXT
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Docetaxel; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (VEGF Trap, Docetaxel) (Experimental): Phase I (closed to accrual as of 3/14/2008): Patients receive VEGF Trap IV over 1 hour on day 1 of course 1. Patients then receive VEGF Trap IV over 1 hour and docetaxel IV over 1 hour on day 1 in all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of VEGF Trap until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 or 6 patients experience dose-limiting toxicity.
  Interventions: Drug: docetaxel; Biological: ziv-aflibercept; Other: laboratory biomarker analysis; Other: pharmacological study
- Phase II Treatment (VEGF Trap, Docetaxel) (Experimental): Phase II (opened to accrual as of 5/9/2008): Patients receive VEGF Trap at the MTD determined in phase I and docetaxel as in phase I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Biological: ziv-aflibercept

INTERVENTIONS:
Drug: docetaxel — 25 mg/m^2 given intravenously (IV) over 1 hour (+/- 10 minutes) following VEGF Trap every 3 weeks starting cycle 1 (21 day cycles)
  Other Names: RP 56976; Taxotere; TXT
Biological: ziv-aflibercept — Starting dose 2 mg/kg given IV Cycle 0. Phase I Group: Every 3 weeks beginning with Cycle 0 (Completed 03/14/2008); Phase II Group: Every 3 weeks starting cycle 1 (Opened 05/09/2008).
  Other Names: aflibercept; vascular endothelial growth factor trap; VEGF Trap; Zaltrap
Other: laboratory biomarker analysis — Correlative studies
  Arms: Treatment (VEGF Trap, Docetaxel)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
  Arms: Treatment (VEGF Trap, Docetaxel)

SUMMARY:
This phase I/II trial is studying the side effects and best dose of VEGF Trap when given together with docetaxel and to see how well they work in treating patients with persistent or recurrent ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer. VEGF Trap may stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving VEGF Trap together with docetaxel may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of VEGF Trap and docetaxel in patients with persistent or recurrent ovarian epithelial, primary peritoneal, or fallopian tube cancer. (Phase I [closed to accrual as of 3/14/2008]) II. Determine the maximum tolerated dose of VEGF Trap in these patients. (Phase I [closed to accrual as of 3/14/2008]) III. Determine the pharmacokinetics of VEGF Trap when administered alone and in combination with docetaxel in these patients. (Phase I [closed to accrual as of 3/14/2008]) IV. Determine the effects of VEGF Trap on tumor perfusion and metabolism in these patients. (Phase I [closed to accrual as of 3/14/2008]) V. Determine the effect of VEGF Trap and docetaxel on circulating endothelial precursors and circulating endothelial cells in these patients. (Phase I [closed to accrual as of 3/14/2008]) VI. Determine the frequency of clinical response (partial response and complete response) in patients treated with this regimen. (Phase II [open to accrual as of 5/9/2008]) VII. Determine the progression-free survival (PFS) and overall survival (OS) of patients treated with this regimen. (Phase II [open to accrual as of 5/9/2008])

SECONDARY OBJECTIVES:

I. Determine the duration of PFS and OS of patients treated with this regimen. (Phase II) II. Determine the frequency and severity of adverse effects of this regimen in these patients. (Phase II) III. Determine the proportion of patients with PFS at 6 months. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of VEGF Trap followed by a phase II study.

PHASE I (closed to accrual as of 3/14/2008): Patients receive VEGF Trap IV over 1 hour on day 1 of course 1. Patients then receive VEGF Trap IV over 1 hour and docetaxel IV over 1 hour on day 1 in all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of VEGF Trap until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 or 6 patients experience dose-limiting toxicity.

PHASE II (opened to accrual as of 5/9/2008): Patients receive VEGF Trap at the MTD determined in phase I and docetaxel as in phase I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients enrolled in phase I (closed to accrual as of 3/14/2008) undergo blood sample collection periodically for pharmacokinetic studies and surrogate marker studies. These patients also undergo dynamic contrast-enhanced MRI, fludeoxyglucose F 18 positron emission tomography, and CT scan at baseline and on day 1 of courses 1 and 2 to evaluate blood flow parameters and metabolic activity of tumors. Patients enrolled in phase I (closed to accrual as of 3/14/2008) and phase II will also undergo blood collection for Anti-VEGF trap antibody.

After the completion of study treatment, patients are followed at 1 and 2 months and then periodically thereafter.

ELIGIBILITY:
Criteria:

* Histologically confirmed ovarian epithelial, primary peritoneal, or fallopian tube cancer:

Persistent or recurrent disease

* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques:

  * Must have >= 1 target lesion to assess response;
  * Tumors within a previously irradiated field are considered nontarget lesions
* Must have received 1 prior platinum-based chemotherapy regimen (for primary disease) containing carboplatin, cisplatin, or other organoplatinum compound:

Initial treatment may have included any of the following:

* High-dose therapy;
* Consolidation therapy;
* Extended therapy administered after surgical or nonsurgical assessment

  * AND Must have received 1 prior platinum-based chemotherapy regimen (for primary disease) containing carboplatin, cisplatin, or other organoplatinum compound:

One additional cytotoxic regimen for recurrent or persistent disease allowed

* No history or evidence of CNS disease, including primary brain tumor or brain metastases
* Zubrod performance status 0-2 (0-1 for patients who received 2 prior regimens [taxane and/or platinum regimens are counted separately])
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* Bilirubin normal
* aspartate aminotransferase / alanine aminotransferase (AST/ALT) < 2.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN OR creatinine clearance > 60 mL/min
* Prothrombin Time (PT)/international normalized ratio (INR) < 1.5 OR in-range INR 2-3 (if patient is on a stable dose of therapeutic warfarin or low molecular weight heparin)
* PTT < 1.2 times control
* Urine protein:creatinine ratio < 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after completion of study treatment
* No active infection requiring antibiotics
* No sensory and motor neuropathy >= grade 2
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to VEGF Trap, Magnevist, or fludeoxyglucose F 18
* No history of allergic reaction to paclitaxel or docetaxel or to products mixed in Cremophor EL or Tween 80
* No active bleeding or pathologic condition that would carry a high risk of bleeding, including any of the following:

Known bleeding disorder; Coagulopathy; Peptic ulcer disease; Diverticulitis; Tumor involving major vessels

* No active and/or untreated pulmonary embolism, deep vein thrombosis, or other thromboembolic event (i.e., any condition associated with aberrant clotting or migration of an induced clot)
* No history or evidence of other CNS disease, including any of the following:

Seizures not controlled with standard medical therapy; Cerebrovascular accident; Transient ischemic attack; Subarachnoid hemorrhage within the past 6 months

* No clinically significant cardiovascular disease, including any of the following:

Uncontrolled hypertension (i.e., systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 100 mm Hg; systolic BP > 180 mm Hg and diastolic BP < 90 mm Hg OR diastolic BP > 90 mm Hg on >= 2 measurements within the past 3 months); Myocardial infarction; Coronary or peripheral artery bypass graft

* No clinically significant cardiovascular disease, including any of the following:

New York Heart association class III or IV congestive heart failure; Serious cardiac arrhythmia requiring medication; Peripheral vascular disease >= grade 2; Unstable angina within the past 6 months; Clinically significant peripheral artery disease (e.g., claudication) within the past 6 months

* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Able to undergo an MRI scan:

No claustrophobia; No implanted devices or metallic foreign bodies not compatible with MRI (e.g., ferromagnetic implants or pacemakers); No known history of allergic reaction to gadolinium contrast agents

* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No significant traumatic injury within the past 28 days
* Recovered from prior therapy to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 grade =< 1:

Alopecia allowed

* No prior VEGF Trap
* No prior cancer treatment that would preclude study treatment
* Prior paclitaxel allowed
* Prior docetaxel for primary or recurrent disease allowed provided the following criteria are met:

No disease progression during therapy; No disease relapse within 3 months of completing therapy; No persistent disease at the completion of primary therapy

* More than 7 days since prior placement of a vascular access device or core biopsy
* At least 1 week since prior hormonal therapy for the malignant tumor
* At least 4 weeks since other prior therapy, including immunologic agents (6 weeks for nitrosoureas or mitomycin C)
* More than 28 days since prior major surgery, open biopsy, dental extraction, or other dental surgery/procedure resulting in an open wound
* No concurrent major surgery
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* No concurrent hematopoietic growth factors during course 1 of phase I
* Concurrent hormone replacement therapy allowed
* White blood count (WBC) >= 3,000/mm^3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coleman, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Derived] Coleman RL, Duska LR, Ramirez PT, Heymach JV, Kamat AA, Modesitt SC, Schmeler KM, Iyer RB, Garcia ME, Miller DL, Jackson EF, Ng CS, Kundra V, Jaffe R, Sood AK. Phase 1-2 study of docetaxel plus aflibercept in patients with recurrent ovarian, primary peritoneal, or fallopian tube cancer. Lancet Oncol. 2011 Nov;12(12):1109-17. doi: 10.1016/S1470-2045(11)70244-3. Epub 2011 Oct 10. PMID 21992853
- See also: The University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 18, 2007 to September 27, 2010. All recruitment done in medical clinic settings.
Pre-assignment Details: Of 58 total participants enrolled at multiple sites, three in the Phase II portion of the study were excluded from the trial.
Groups:
- Phase I VEGF Trap, Docetaxel: Phase I VEGF Trap starting dose 2 mg/kg intravenous (IV) over 1 hour on day 1 of course 1, then VEGF Trap IV and Docetaxel 75 mg/m^2 IV over 1 hour on day 1 in all subsequent courses. Courses repeat every 21 days. Escalating doses of VEGF Trap (2, 4, or 6 mg/kg) until maximum tolerated dose (MTD) determined.
- Phase II: VEGF Trap, Docetaxel: Phase II VEGF Trap 6 mg/kg (the MTD determined in Phase I) and Docetaxel 75 mg/m^2 as in Phase I. Courses repeat every 21 days.
Period: Complete Study Participation
Arm/Group | Phase I VEGF Trap, Docetaxel | Phase II: VEGF Trap, Docetaxel
Started | 9 (Phase 1 opened on January 17, 2007 and closed to new patient entry on March 7, 2008.) | 49 (After toxicity observations, Phase 2 opened June 4, 2008 and closed September 27, 2010.)
Completed | 9 | 49
Not Completed | 0 | 0
Period: Phase 1: VEGF Trap Escalating Dose
Arm/Group | Phase I VEGF Trap, Docetaxel | Phase II: VEGF Trap, Docetaxel
Started | 9 (Phase 1 opened on January 17, 2007 and closed to new patient entry on March 7, 2008.) | 0 (Participants registered in next period.)
Completed | 9 | 0
Not Completed | 0 | 0
Period: Phase 2: MTD VEGF Trap + Docetaxel
Arm/Group | Phase I VEGF Trap, Docetaxel | Phase II: VEGF Trap, Docetaxel
Started | 0 | 49 (After toxicity observations Phase 2 opened June 4, 2008 and closed to entry September 27, 2010.)
Completed | 0 | 46
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Incomplete Assessment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase II VEGF Trap, Docetaxel: Phase II VEGF Trap 6 mg/kg (the MTD determined in Phase I) and Docetaxel 75 mg/m^2 as in Phase I. Courses repeat every 21 days.
- Total: Total of all reporting groups
Arm/Group | Phase I VEGF Trap, Docetaxel | Phase II VEGF Trap, Docetaxel | Total
Number analyzed (Participants) | 9 | 46 | 55
Age, Continuous [Median (Full Range); unit: years] | 59 [49 to 71] | 58 [38 to 80] | 58 [38 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 46 | 55
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 44 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 45 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 46 | 55
Participant Cancer Histology [Number; unit: participants] — Histological classification of participant cancer based on pathology report from most recent pre-registration diagnostic biopsy or surgery, confirmed within 14 days after registration for baseline measurements/data.
  participants
    Adenocarcinoma | 0 | 3 | 3
    Clear cell | 1 | 4 | 5
    Endometrioid | 0 | 1 | 1
    Mixed | 0 | 5 | 5
    Serous | 6 | 31 | 37
    Transitional cell | 2 | 0 | 2
    Unclassified | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of VEGF Trap (Phase I)
Description: Escalating dose levels of VEGF Trap were administered intravenously over three dose levels (2, 4, or 6 mg/kg; one dose every 21 days) to identify the maximum tolerated dose (MTD). The MTD is defined as the highest dose level below which 2 or more patients encounter a dose limiting toxicity (DLT), graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. MTD established on absence of observed DLT(s) in either cycle 0 (single agent) or cycle 1 (combination therapy) of any given dose level.
Time Frame: 21 day cycle, up to 3 cycles
Measure: Number; unit: mg/kg
Arm/Group | Phase I VEGF Trap, Docetaxel
Number analyzed (Participants) | 9
mg/kg | 6

2. Primary Outcome: Number of Participants With Clinical Response (Partial Response or Complete Response) According to the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Frequency of clinical response (partial response or complete response) according to the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR): Disappearance all target lesions; Partial Response (PR): >/= 30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD; Progressive Disease (PD): >/= 20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of 1+ new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum LD since treatment started.
Time Frame: Up to 6 months
Measure: Number; unit: participants
Arm/Group | Phase I VEGF Trap, Docetaxel | Phase II: VEGF Trap, Docetaxel
Number analyzed (Participants) | 9 | 46
participants
  Complete Response | 0 | 11
  Partial Response | 2 | 14

3. Primary Outcome: Median Overall Survival (OS) (Phase II)
Description: Overall survival was defined from the date of study entry until death or date of last contact. Median survival time points calculated in the method of Kaplan-Meier. Standard RECIST criteria followed to evaluate response and progression, and all documented responses required confirmation by imaging, examination, or both, no sooner than 4 weeks after the initial documentation of response. In the absence of new symptoms, response assessment consistently done after two additional cycles of therapy.
Time Frame: Time from start of treatment to time of progression, assessed up to 6 years.
Measure: Median (Full Range); unit: months
Arm/Group | Phase II: VEGF Trap, Docetaxel
Number analyzed (Participants) | 46
months | 26.6 [13.1 to 49.5]

4. Primary Outcome: Overall Objective Response Rate According to RECIST (Phase II)
Description: The percentage of participants in the Phase II arm with an objective response defined as a measurable response according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. Standard RECIST criteria were followed to evaluate response and progression. All documented responses were required to undergo confirmation by imaging, examination, or both, no sooner than 4 weeks after the initial documentation of response. In the absence of new symptoms, this response assessment was consistently done after two additional cycles of therapy.
Time Frame: Up to 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: VEGF Trap, Docetaxel
Number analyzed (Participants) | 46
percentage of participants | 54

5. Primary Outcome: Median Progression-Free Survival (PFS) (Phase II)
Description: Progression-Free Survival was calculated from study entry until documented disease, death or date of last contact.
Time Frame: Time from start of treatment to time of progression, assessed up to 6 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: VEGF Trap, Docetaxel
Number analyzed (Participants) | 46
months | 6.4 [5.1 to 10.3]

6. Secondary Outcome: Overall Median Duration of Response (Phase II)
Description: Duration of the response from time response is achieved until disease progression is detected. Response assessed following treatment (every 3 weeks) for disease progression. Study duration January 2007 to May 2013, approximately six and half years.
Time Frame: Response assessed following treatment (every 3 weeks), up to 6 years. Study duration January 2007 to May 2013.
Population: Number analyzed represents those Phase II participants with response as documented in Outcome Measure 2.
Measure: Median (Full Range); unit: months
Arm/Group | Phase II: VEGF Trap, Docetaxel
Number analyzed (Participants) | 25
months | 6.0 [1.8 to 27.0]

7. Secondary Outcome: Number of Participants With Treatment-related Adverse Effects as Assessed by NCI CTCAE v3.0 (Phase II)
Description: Number of participants with adverse effects of treatment. Frequency and severity of adverse effects of treatment as assessed by NCI CTCAE v3.0 (Phase II)
Time Frame: Up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I VEGF Trap, Docetaxel | Phase II: VEGF Trap, Docetaxel
Number analyzed (Participants) | 9 | 49
Participants | 9 | 46

8. Secondary Outcome: Number of Participants With PFS (Phase II)
Description: Progression-free survival (PFS) defined as number of participants out of total in arm that had no disease progression as measured at 6 months. Standard RECIST criteria used to evaluate response and progression. All documented responses required confirmation by imaging, examination, or both, no sooner than 4 weeks after initial documentation of response. In the absence of new symptoms, response assessment was consistently done after two additional cycles of therapy.
Time Frame: 6 months
Population: Phase I, 2 participants had partial response and 3 were stable disease for a total of 5 responses but only 2 had a Clinical Response (confirmed).
  Phase II, 46 participants was evaluable out of 49 enrolled for response/toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I VEGF Trap, Docetaxel | Phase II: VEGF Trap, Docetaxel
Number analyzed (Participants) | 9 | 46
Participants
  Partial Response | 2 | 11
  No change/Stable Disease | 3 | 10
  Progressive Disease | 4 | 14
  Complete Response | 0 | 11

ADVERSE EVENTS:
Time Frame: Adverse events that occur up to 30 days after the last dose of treatment were collected. Among all Phase 2 participants, 307 treatment cycles of 21 days were administered (median 6, range 1-22).
Arm/Group | Phase I VEGF Trap, Docetaxel | Phase II: VEGF Trap, Docetaxel
Serious Adverse Events (participants affected / at risk) | 8/9 | 43/46
Other Adverse Events (participants affected / at risk) | 9/9 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I VEGF Trap, Docetaxel (N=9) | Phase II: VEGF Trap, Docetaxel (N=46)
Lowered leucocytes (Blood and lymphatic system disorders) | 4 | 25
Neutropenia (Blood and lymphatic system disorders) | 8 | 37
Prolonged PTT (Blood and lymphatic system disorders) | 1 | 0
Lowered magnesium (Metabolism and nutrition disorders) | 0 | 1
Raised creatinine (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Cardiac disorders) | 2 | 0
Fatigue (General disorders) | 4 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Neuropathy, sensory (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3
Headache (General disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I VEGF Trap, Docetaxel (N=9) | Phase II: VEGF Trap, Docetaxel (N=46)
Lowered haemoglobin (Blood and lymphatic system disorders) | 4 | 19
Lowered platelets (Blood and lymphatic system disorders) | 4 | 12
Lowered leucocytes (Blood and lymphatic system disorders) | 5 | 13
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Prolonged PTT (Blood and lymphatic system disorders) | 2 | 3
Lowered magnesium (Metabolism and nutrition disorders) | 3 | 19
Lowered potassium (Metabolism and nutrition disorders) | 2 | 4
Raised Alanine transaminase (ALT) (Metabolism and nutrition disorders) | 1 | 4
Raised Aspartate aminotransferase (AST) (Metabolism and nutrition disorders) | 4 | 7
Raised alkaline phosphatase (Metabolism and nutrition disorders) | 0 | 11
Raised creatinine (Metabolism and nutrition disorders) | 0 | 5
Hypertension (Cardiac disorders) | 5 | 5
Fatigue (General disorders) | 5 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 20
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 10
Infection, nail beds (Skin and subcutaneous tissue disorders) | 0 | 5
Watery eyes (Eye disorders) | 1 | 22
Voice changes (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Infection (Infections and infestations) | 3 | 5
Neuropathy, sensory (Nervous system disorders) | 2 | 17
Hand or foot reaction (Skin and subcutaneous tissue disorders) | 2 | 6
Nose bleeds (Respiratory, thoracic and mediastinal disorders) | 4 | 22
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 35
Stomatitis (Gastrointestinal disorders) | 8 | 33
Headache (General disorders) | 6 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less